CLINICAL TRIAL: NCT01364597
Title: Open-label, Single-arm, Multicenter, Long-term Study to Evaluate Safety and Efficacy of Brivaracetam Used as Adjunctive Treatment in Pediatric Subjects With Epilepsy
Brief Title: Open-label Long-term Study of Adjunctive Brivaracetam in Pediatric Subjects With Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01266; 2011-000374-60 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Results first posted 2022-08-29 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy
Keywords: Brivaracetam; Epilepsy; Child; Infant; Adolescents; Partial onset seizures
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brivaracetam (Experimental)
  Interventions: Drug: Brivaracetam (BRV)

INTERVENTIONS:
Drug: Brivaracetam (BRV) — The max BRV dose will be 5.0 mg/kg/day, not to exceed a dose of 200 mg/day for subjects with body weight >40kg. Subjects may receive oral solution or oral tablets. The LTFU subjects will start dosing in N01266 on the individualized BRV dose they were receiving at the completion of the core study. Subjects must be able to tolerate the min BRV dose specified in the core study to be eligible for entry into the Evaluation Period of N01266. Dose can be adjusted as considered necessary by the Investigator and required by the subject's medical condition. All subjects who prematurely discontinue the study should complete an EDV and have their BRV dose down titrated by a maximum of half the dose every week for a maximum of 4 weeks until a dose of 1 mg/kg/day (50 mg/day for subjects with body weights >50kg) is reached.

SUMMARY:
This study will evaluate the safety and tolerability of brivaracetam in pediatric subjects with epilepsy.

DETAILED DESCRIPTION:
This is a Phase 3, open-label, single-arm, multicenter, long-term study to evaluate the safety and efficacy of brivaracetam (BRV) in children with epilepsy.

This study was initially designed for pediatric subjects who had completed a previous BRV study.

With protocol amendment 4, enrollment for "directly enrolled" subjects was modified from 'up to' an additional 100 subjects to "at least" 100 subjects, keeping the planned total enrollment of approximately 600 subjects to allow flexibility in the number of patients reaching 1 year of exposure.

With protocol amendment 5, entry criteria for subjects coming for other pediatric core studies in development were included. Additional clarity was provided for subjects enrolled in N01266 that temporary roll over to one of those studies and resume participation in N01266.

With protocol amendment 6, central EEG reading and entry visit EEG were removed. Some clarifications on study assessments (questionnaires, EEGs) was provided and inclusion criteria were aligned from an earlier local amendment.

With protocol amendment 7, the pregnancy section was updated to clarify that Pregnancy Report and Outcome Form has to be completed in all pregnancies.

With protocol amendment 8, re-categorization of study variables in compliance with reporting registries was performed. Modifications due to COVID19 pandemic were implemented and clarification provided that participants may transition to another BRV study.

The primary objective is to evaluate the long-term safety and tolerability of BRV. The secondary objective is to assess the efficacy of BRV during long-term exposure.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

* Informed Consent form (ICF) is signed and dated by the parent(s) or legal representative(s)
* Subject/legal representative is considered reliable and capable of adhering to the protocol
* For female subjects:
* Subject is not of childbearing potential

OR if women of childbearing potential, and sexually active only if:

* Adequate Contraceptive method
* Negative pregnancy test
* Understands the consequences and potential risks of inadequately protected sexual activity, understands and properly uses contraceptive methods, and is willing to inform the Investigator of any contraception changes

Long Term Follow-up Subjects:

- Male or female subjects having participated in a core study with a confirmed diagnosis of epilepsy and for whom a reasonable benefit from long-term administration of BRV is expected

Directly Enrolled Subjects:

* Subject is a male or female ≥4 years to <17 years of age
* Subject has a clinical diagnosis of partial-onset seizures (POS) according to the International League Against Epilepsy (ILAE) classification
* Subject has an EEG compatible with the clinical diagnosis of POS
* Subject has been observed to have uncontrolled POS after an adequate course of treatment (in the opinion of the Investigator) with at least 1 antiepileptic drug (AED; concurrently or sequentially)
* Subject had at least 1 seizure (POS) during the 3 weeks before the Screening Visit (ScrV)
* Subject is taking at least 1 AED. All AEDs need to be at a stable dose for at least 7 days before the ScrV. Vagal nerve stimulator stable for at least 2 weeks before the ScrV is allowed and will be counted as a concomitant AED. Benzodiazepines taken more than once a week (for any indication) will be considered as a concomitant AED

Exclusion Criteria:

All Subjects:

* Subject is a pregnant or nursing female
* Subject has severe medical, neurological, or psychiatric disorders or laboratory values, which may have an impact on the safety of the subject.
* Subject has planned participation in any clinical study of another investigational drug or device.
* Subject has >1.5x upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >1.0xULN total bilirubin (≥1.5xULN total bilirubin if known Gilbert's syndrome). If subject has elevations only in total bilirubin that are >ULN and <1.5xULN, fractionate bilirubin to identify possible undiagnosed Gilbert's syndrome (ie, direct bilirubin <35%). N01349 subjects with a total bilirubin > ULN may be considered for the study if benign unconjugated hyperbilirubinemia is suspected in the context of prolonged neonatal jaundice, after discussion with the medical monitor. For randomized subjects with a baseline result >ULN for ALT, AST, ALP, or total bilirubin, a baseline diagnosis and/or the cause of any clinically meaningful elevation must be understood and recorded in the eCRF. If subject has >ULN ALT, AST, or ALP that does not meet the exclusion limit at the baseline referenced in Table 5-1 for LTFU subjects and at the Screening Visit for directly enrolled subjects, repeat the tests, if possible, prior to dosing to ensure there is no further ongoing clinically relevant increase. In case of a clinically relevant increase, inclusion of the subject must be discussed with the Medical Monitor. Tests that result in ALT, AST, or ALP up to 25% above the exclusion limit may be repeated once for confirmation. This includes re-screening.
* Subject has chronic liver disease.

Long Term Follow-up Subjects:

* Subject had hypersensitivity to BRV or excipients or comparative drugs as stated in this protocol during the course of the core study.
* Subject had poor compliance with the visit schedule or medication intake in the core study.
* Subject ≥6 years of age has a lifetime history of suicide attempt (including actual attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at the EV. If a subject has active suicidal ideation without a specific plan as indicated by a positive response ("Yes") to Question 4 of Columbia-Suicide Severity Rating Scale (C SSRS) at the EV, the subject should be referred immediately to a Mental Healthcare Professional and may be excluded from the study based upon the Investigator's judgment of benefit/risk of continuing the subject in the study/on study medication.

Directly Enrolled Subjects:

* Subject has previously received BRV.
* Subject had concomitant use of LEV at the ScrV. In addition, the use of LEV is prohibited for at least 4 weeks prior to the ScrV.
* Subject has epilepsy secondary to a progressive cerebral disease or tumor, or any other progressively neurodegenerative disease. Stable arteriovenous malformations, meningiomas or other benign tumors may be acceptable according to Investigator's opinion.
* Subject has a history of primary generalized epilepsy.
* Subject has a history of status epilepticus in the month immediately prior to the ScrV or during the Up Titration Period.
* Subject has a history or presence of pseudoseizures.
* Subject is suffering only from febrile seizures.
* Subject is on felbamate with less than 18 months continuous exposure. Subject who has taken felbamate for a combined duration of treatment and wash out of <18 months before the ScrV.
* Subjects treated with vigabatrin who have visual field defects.
* Subject has an allergy to pyrrolidone derivatives or investigational product excipients or a history of multiple drug allergies.
* Subject has any clinically significant acute or chronic illness as determined during the physical examination or from other information available to the Investigator (eg, bone marrow depression, chronic hepatic disease, severe renal impairment, psychiatric disorder).
* Subject has an underlying disease or is receiving a treatment that may interfere with the absorption, distribution, metabolism, and elimination of the study drug.
* Subject has any medical condition that might interfere with his/her study participation (eg, serious infection or scheduled elective surgery).
* Subject has a terminal illness.
* Subject has any clinically significant deviations from reference range values for laboratory parameters as determined by the Investigator.
* Subject has a clinically relevant ECG abnormality according to the Investigator.
* Subject had major surgery within 6 months prior to the ScrV.
* Subject received any investigational drug or device within the 30 days prior to the ScrV.

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 257 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 877 822 9493 (UCB)
Locations (56):
- United States (15):
  - N01266 243, Los Angeles, California
  - N01266 108, Gulf Breeze, Florida
  - N01266 103, Wellington, Florida
  - N01266 118, Chicago, Illinois
  - N01266 106, Boston, Massachusetts
  - N01266 101, Saint Paul, Minnesota
  - N01266 113, Chesterfield, Missouri
  - N01266 105, Buffalo, New York
  - N01266 252, New York, New York
  - N01266 104, Rochester, New York
  - N01266 237, Durham, North Carolina
  - N01266 107, Cincinnati, Ohio
  - N01266 111, Columbus, Ohio
  - N01266 114, Pittsburgh, Pennsylvania
  - N01266 117, Houston, Texas
- Belgium (4):
  - N01266 202, Brussels
  - N01266 203, Brussels
  - N01266 201, Leuven
  - N01266 204, Leuven
- Czechia (3):
  - N01266 502, Hradec Králové
  - N01266 504, Ostrava Prouba
  - N01266 240, Prague
- France (2):
  - N01266 207, Lille
  - N01266 206, Paris
- Germany (2):
  - N01266 218, Bayern
  - N01266 209, Freiburg im Breisgau
- Hungary (5):
  - N01266 210, Budapest
  - N01266 224, Budapest
  - N01266 247, Budapest
  - N01266 222, Debrecen
  - N01266 232, Miskolc
- N01266 211, Cork, Ireland
- Italy (6):
  - N01266 212, Messina
  - N01266 213, Parma
  - N01266 238, Pavia
  - N01266 239, Pavia
  - N01266 230, Roma
  - N01266 256, Roma
- Mexico (5):
  - N01266 223, Aguascalientes
  - N01266 611, Chihuahua City
  - N01266 609, Culiacán
  - N01266 603, Guadalajara
  - N01266 610, Monterrey
- Poland (7):
  - N01266 404, Bialystok
  - N01266 403, Gdansk
  - N01266 406, Kielce
  - N01266 402, Krakow
  - N01266 401, Poznan
  - N01266 407, Szczecin
  - N01266 405, Wroclaw
- Spain (5):
  - N01266 309, Barcelona
  - N01266 306, Madrid
  - N01266 301, Palma de Mallorca
  - N01266 248, Seville
  - N01266 308, Valencia
- N01266 215, London, United Kingdom

REFERENCES:
- [Result] Lagae L, Klotz KA, Fogarasi A, Floricel F, Reichel C, Elshoff JP, Fleyshman S, Kang H. Long-term safety and efficacy of adjunctive brivaracetam in pediatric patients with epilepsy: An open-label, follow-up trial. Epilepsia. 2023 Nov;64(11):2934-2946. doi: 10.1111/epi.17754. Epub 2023 Sep 5. PMID 37597326
- [Result] Bourikas D, Elmoufti S, Elshoff JP, Little A, Pucylowski K, Moseley B, Lagae L. Long-term tolerability and efficacy of adjunctive brivaracetam in pediatric patients with generalized-onset seizures: Subgroup analysis of an open-label, follow-up trial. Epilepsy Behav. 2025 Oct;171:110569. doi: 10.1016/j.yebeh.2025.110569. Epub 2025 Jul 29. PMID 40737960
- [Derived] Markham A. Brivaracetam: First Global Approval. Drugs. 2016 Mar;76(4):517-22. doi: 10.1007/s40265-016-0555-6. PMID 26899665
- See also: Product Information — http://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in August 2011 and concluded in February 2022.
Pre-assignment Details: The Participant Flow refers to the Enrolled Set.
Groups:
- Age Cohort: ≥1 Month to <2 Years: Participants from core study (LTFU [Long term follow-up] participants from N01263 [NCT00422422], EP0065 [NCT03405714] or N01349 [NCT03325439]) aged greater than or equal to (≥) 1 month to less than (<) 2 years entered evaluation period (EP) and received individualized Brivaracetam (BRV) dose as they were receiving at completion of core study. For all participants, the approximate BRV doses to be administered are 1 to 5 milligrams per kilogram per day (mg/kg/day) (0.5, 1, 2, and 2.5 mg/kg twice daily[bid]), tablet or oral solution and can be up-titrated or down-titrated based on investigator decision with a maximum allowable BRV dose of 5.0 mg/kg/day (2.5 mg/kg bid), not to exceed a dose of 200 mg/day. The duration of the treatment for each participant was planned to be at least 3 years, until BRV received approval for pediatric participants in their age range or until the investigational medicinal product (IMP) development was stopped by the Sponsor.
- Age Cohort: ≥2 to <4 Years: Participants from core study (LTFU participants from N01263 [NCT00422422] and EP0065 [NCT03405714]) aged ≥2 Years to <4 years entered EP and received individualized BRV dose as they were receiving at completion of core study. For all participants, the approximate BRV doses to be administered are 1 to 5 mg/kg/day (0.5, 1, 2, and 2.5mg/kg bid), tablet or oral solution and can be up-titrated or down-titrated based on investigator decision with a maximum allowable BRV dose of 5.0 mg/kg/day (2.5mg/kg bid), not to exceed a dose of 200mg/day. The duration of the treatment for each participant was planned to be at least 3 years, until BRV received approval for pediatric participants in their age range or until the IMP development was stopped by the Sponsor.
- Age Cohort: ≥4 to <12 Years: Participants from core study (LTFU participants from N01263 [NCT00422422] and EP0065 [NCT03405714]) aged ≥4 Years to <12 years entered EP and received individualized BRV dose as they were receiving at completion of core study and Directly Enrolled (DE) participants in this study aged ≥4 years to <12 years of age received BRV dose based on tolerability confirmed during screening period. For all participants, the approximate BRV doses to be administered are 1 to 5 mg/kg/day (0.5, 1, 2, and 2.5mg/kg bid), tablet or oral solution and can be up-titrated or down-titrated based on investigator decision with a maximum allowable BRV dose of 5.0 mg/kg/day (2.5 mg/kg bid), not to exceed a dose of 200 mg/day. The duration of the treatment for each participant was planned to be at least 3 years, until BRV received approval for pediatric participants in their age range or until the IMP development was stopped by the Sponsor.
- Age Cohort: ≥12 to <17 Years: Participants from core study (LTFU participants from N01263 [NCT00422422] and EP0065 [NCT03405714]) aged ≥12 Years to <17 years entered EP and received individualized BRV dose as they were receiving at completion of core study and DE participants in this study aged ≥12 years to <17 years of age received BRV dose based on tolerability confirmed during screening period. For all participants, the approximate BRV doses to be administered are 1 to 5 mg/kg/day (0.5, 1, 2, and 2.5 mg/kg bid), tablet or oral solution and can be up-titrated or down-titrated based on investigator decision with a maximum allowable BRV dose of 5.0 mg/kg/day (2.5 mg/kg bid), not to exceed a dose of 200 mg/day. The duration of the treatment for each participant was planned to be at least 3 years, until BRV received approval for pediatric participants in their age range or until the IMP development was stopped by the Sponsor.
Period: Overall Study
Arm/Group | Age Cohort: ≥1 Month to <2 Years | Age Cohort: ≥2 to <4 Years | Age Cohort: ≥4 to <12 Years | Age Cohort: ≥12 to <17 Years
Started | 36 | 15 | 141 | 65
Directly Enrolled (DE) Participants | 0 | 0 | 85 | 35
Long-term Follow-up (LTFU) Participants | 36 | 15 | 56 | 30
Completed | 18 | 4 | 65 | 37
Not Completed | 18 | 11 | 76 | 28
Not completed — Adverse Event | 4 | 5 | 16 | 7
Not completed — Lack of Efficacy | 4 | 4 | 23 | 8
Not completed — Protocol Violation | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 5 | 3
Not completed — Withdrawal by Subject | 4 | 1 | 18 | 6
Not completed — Non compliance | 1 | 0 | 1 | 0
Not completed — Lack of compliance | 1 | 0 | 0 | 0
Not completed — End of treatment epilepsy | 1 | 0 | 0 | 0
Not completed — No Seizures | 1 | 0 | 0 | 0
Not completed — Lack of reliability from the subject's caregiver | 1 | 0 | 0 | 0
Not completed — Cure | 1 | 0 | 0 | 0
Not completed — Patient was moving | 0 | 1 | 0 | 0
Not completed — Seizures resolved | 0 | 0 | 1 | 0
Not completed — Patient became seizure-free after surgery | 0 | 0 | 1 | 0
Not completed — 5 year without seizures. Treatment is finish | 0 | 0 | 1 | 0
Not completed — Patient cured from Epilepsy | 0 | 0 | 1 | 0
Not completed — Investigator decision | 0 | 0 | 1 | 0
Not completed — Sponsor recommended discontinuation | 0 | 0 | 0 | 1
Not completed — Parents went abroad with the patient | 0 | 0 | 1 | 0
Not completed — BRV discontinued as no seizures during 2 years | 0 | 0 | 1 | 0
Not completed — BRV administration dropout | 0 | 0 | 1 | 0
Not completed — Dropout | 0 | 0 | 3 | 1
Not completed — Unreliable subject | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refers to the Enrolled Set (ES) which included all study participants with epilepsy who gave informed consent, or for whom informed consent was given by parent(s)/legal representative(s).
Groups:
- Total: Total of all reporting groups
Arm/Group | Age Cohort: ≥1 Month to <2 Years | Age Cohort: ≥2 to <4 Years | Age Cohort: ≥4 to <12 Years | Age Cohort: ≥12 to <17 Years | Total
Number analyzed (Participants) | 36 | 15 | 141 | 65 | 257
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36 | 15 | 141 | 65 | 257
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.122 (0.504) | 2.761 (0.582) | 7.699 (2.394) | 13.824 (1.274) | 8.039 (4.529)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 5 | 62 | 30 | 116
  Male | 17 | 10 | 79 | 35 | 141
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/ Alaskan native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Black | 0 | 0 | 2 | 2 | 4
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 28 | 14 | 107 | 48 | 197
  Other/Mixed | 8 | 1 | 32 | 15 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 1 | 38 | 19 | 69
  Not Hispanic or Latino | 24 | 14 | 103 | 46 | 187
  Missing | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) During the Study
Description: TEAEs are defined as AEs that had onset on or after the day of first BRV dose.
Time Frame: From Baseline to end of study (up to 10 years)
Population: The Safety Set (SS) consisted of all enrolled participants who took at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Age Cohort: ≥1 Month to <2 Years | Age Cohort: ≥2 to <4 Years | Age Cohort: ≥4 to <12 Years | Age Cohort: ≥12 to <17 Years
Number analyzed (Participants) | 36 | 15 | 141 | 65
percentage of participants | 94.4 | 93.3 | 93.6 | 92.3

2. Primary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (SAEs) During the Study
Description: TEAEs are defined as AEs that had onset on or after the day of first BRV dose. A SAE was defined as an event that met 1 or more of the below criteria: a) Death, b) Life-threatening, (Life-threatening did not include a reaction that might have caused death had it occurred in a more severe form.) c) Significant or persistent disability/incapacity, d) Congenital anomaly/birth defect (including that occurring in a fetus), e) Important medical event that, based upon appropriate medical judgment, may have jeopardized participant and may have required medical or surgical intervention to prevent 1 of the other outcomes listed in the definition of serious, (Important medical events may have included allergic bronchospasm requiring intensive treatment in an emergency room [ER] or at home) f) Initial inpatient hospitalization or prolongation of hospitalization. (A participant admitted to a hospital, even if released on the same day, met the criteria for the initial inpatient hospitalization).
Time Frame: From Baseline to end of study (up to 10 years)
Population: The Safety Set (SS) consisted of all enrolled participants who took at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Age Cohort: ≥1 Month to <2 Years | Age Cohort: ≥2 to <4 Years | Age Cohort: ≥4 to <12 Years | Age Cohort: ≥12 to <17 Years
Number analyzed (Participants) | 36 | 15 | 141 | 65
percentage of participants | 38.9 | 53.3 | 29.8 | 29.2

3. Secondary Outcome: Absolute Change in 28-days Adjusted Partial-onset-seizure (POS) Frequency for Participants Aged ≥2 Years From Baseline to the End of the Evaluation Period in Participants With POS Only (Based on Daily Record Card [DRC])
Description: Absolute change in seizure frequency per 28 days based on the daily record card (DRC) data, is calculated as baseline seizure frequency per 28 days minus post-Baseline seizure frequency per 28 days. The 28 day adjusted seizure frequency was calculated by dividing the number of partial seizures by the number of days for which the diary was completed, and multiplying the resulting value by 28. This OM was analyzed in participants ≥2 years (per DRC data) only.
  Here in the study FAS indicates Full Analysis Set, EEG indicates electroencephalogram, OM indicates Outcome measure
Time Frame: From Baseline (LTFU participants: Baseline of previous studies N01263 [NCT00422422]; and DE participants: Baseline of current study) to the end of the evaluation period (up to 10 years)
Population: FAS: enrolled participants who had at least 1 dose of study drug in the study and had at least 1 completed post-baseline DRC or EEG. Overall number of participants analyzed consist of all participants (≥2 years only [per DRC data]) evaluable for this OM and it differs in absolute and percent change OMs as later cannot be analyzed with 0 baseline ADF. Per plan, participants were grouped per cohort linked to source (DRC for ≥2 years/EEG for <2 years) from which their seizure data is recorded.
Measure: Mean (Standard Deviation); unit: seizure frequency per 28-days
Groups:
- Brivaracetam (BRV): Participants ≥ 2 Years to <17 Years: Participants from core study (LTFU participants from N01263 [NCT00422422]) aged ≥2 Years to <17 years entered EP and received individualized BRV dose as they were receiving at completion of core study and DE participants in this study aged ≥4 years to <17 years of age received BRV dose based on tolerability confirmed during screening period. For all participants, the approximate BRV doses to be administered are 1 to 5 mg/kg/day (0.5, 1, 2, and 2.5 mg/kg bid), tablet or oral solution and can be up-titrated or down-titrated based on investigator decision with a maximum allowable BRV dose of 5.0 mg/kg/day (2.5 mg/kg bid), not to exceed a dose of 200 mg/day. The duration of the treatment for each participant was planned to be at least 3 years, until BRV received approval for pediatric participants in their age range or until the IMP development was stopped by the Sponsor.
Arm/Group | Brivaracetam (BRV): Participants ≥ 2 Years to <17 Years
Number analyzed (Participants) | 134
seizure frequency per 28-days | -37.48 (628.34)

4. Secondary Outcome: Percent Change in 28-days Adjusted Partial-onset-seizure (POS) Frequency for Participants Aged ≥2 Years From Baseline to the End of the Evaluation Period in Participants With POS Only (Based on DRC Data)
Description: Percent change is calculated as absolute change in seizure frequency per 28 days divided by baseline seizure frequency per 28 Days multiplied to 100. The 28 day adjusted seizure frequency was calculated by dividing the number of partial seizures by the number of days for which the diary was completed, and multiplying the resulting value by 28. This OM was analyzed in participants ≥2 years (per DRC data) only.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Brivaracetam (BRV): Participants ≥ 2 Years to <17 Years
Number analyzed (Participants) | 105
percent change | 26.57 (123.06)

5. Secondary Outcome: 50% Responder Rate for Participants ≥2 Years of Age for Total Seizures (All Types) (Based on DRC Data)
Description: A responder is defined as a participant with a ≥50% reduction in seizure frequency from the baseline period of the previous study for LTFU participants or during this study for DE participants. This OM was analyzed in participants ≥2 years (per DRC data) only.
Time Frame: as for outcome 3
Population: FAS: all enrolled participants who took at least 1 dose of study drug in this Long-term study and had at least 1 completed post-baseline DRC or EEG. Overall number of participants analyzed included all participants evaluable for this OM. Per planned analysis, participants were grouped as per cohort linked to source (DRC for ≥2 years /EEG for <2 years) from which their seizure data is recorded. This OM was analyzed in participants ≥2 years of age (per DRC data) only.
Measure: Number; unit: percentage of participants
Groups:
- Brivaracetam (BRV): Participants ≥2 Years to <17 Years: Participants from core study (LTFU participants from N01263 [NCT00422422]) aged ≥2 Years to <17 years entered EP and received individualized BRV dose as they were receiving at completion of core study and DE participants in this study aged ≥4 years to <17 years of age received BRV dose based on tolerability confirmed during screening period. For all participants, the approximate BRV doses to be administered are 1 to 5 mg/kg/day (0.5, 1, 2, and 2.5 mg/kg bid), tablet or oral solution and can be up-titrated or down-titrated based on investigator decision with a maximum allowable BRV dose of 5.0 mg/kg/day (2.5 mg/kg bid), not to exceed a dose of 200 mg/day. The duration of the treatment for each participant was planned to be at least 3 years, until BRV received approval for pediatric participants in their age range or until the IMP development was stopped by the Sponsor.
Arm/Group | Brivaracetam (BRV): Participants ≥2 Years to <17 Years
Number analyzed (Participants) | 167
percentage of participants | 50.9

6. Secondary Outcome: Absolute Change in Average Daily Frequency (ADF) of Partial-onset-seizures (POS) in Participants <2 Years of Age With POS Only (Based on EEG Data)
Description: Absolute change in ADF is calculated as the baseline ADF minus post-baseline ADF. ADF is calculated as (number of seizures from central reader divided by stop date and time of EEG minus start date and time of EEG) multiplied to 60, multiplied to 24. This OM was analyzed in participants <2 years (per EEG data) only.
Time Frame: From Baseline (LTFU participants: Baseline of previous studies N01263 [NCT00422422] or N01349 [NCT03325439]) to the end of the evaluation period (up to 10 years)
Population: FAS: enrolled participants who had at least 1 dose of study drug in the study and had at least 1 completed post-baseline DRC or EEG. Overall number of participants analyzed consist of all participants (<2 years only [per EEG data]) evaluable for this OM and it differs in absolute and percent change OMs as later cannot be analyzed with 0 baseline ADF. Per plan, participants were grouped per cohort linked to source (DRC for ≥2 years/EEG for <2 years) from which their seizure data is recorded.
Measure: Mean (Standard Deviation); unit: seizures per day
Groups:
- Brivaracetam (BRV): Participants ≥1 Month to <2 Years: Participants from core study (LTFU [Long term follow-up] participants from N01263 [NCT00422422] or N01349 [NCT03325439]) aged ≥1 month to <2 years entered EP and received individualized BRV dose as they were receiving at completion of core study. For all participants, the approximate BRV doses to be administered are 1 to 5 mg/kg/day (0.5, 1, 2, and 2.5 mg/kg bid), tablet or oral solution and can be up-titrated or down-titrated based on investigator decision with a maximum allowable BRV dose of 5.0 mg/kg/day (2.5 mg/kg bid), not to exceed a dose of 200 mg/day. The duration of the treatment for each participant was planned to be at least 3 years, until BRV received approval for pediatric participants in their age range or until the IMP development was stopped by the Sponsor.
Arm/Group | Brivaracetam (BRV): Participants ≥1 Month to <2 Years
Number analyzed (Participants) | 8
seizures per day | 2.56 (4.44)

7. Secondary Outcome: Percent Change in Average Daily Frequency (ADF) of Partial-onset-seizures (POS) in Participants <2 Years of Age With POS Only (Based on EEG Data)
Description: Percent change in average daily frequency (ADF) is calculated as absolute change in ADF divided by baseline ADF multiplied to 100. ADF is calculated as (number of seizures from central reader divided by stop date and time of EEG minus start date and time of EEG) multiplied to 60, multiplied to 24. This OM was analyzed in participants <2 years (per EEG data) only.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Brivaracetam (BRV): Participants ≥1 Month to <2 Years
Number analyzed (Participants) | 3
percent change | 98.72 (2.22)

8. Secondary Outcome: 50% Responder Rate for Participants <2 Years of Age for Total Seizures (All Types) (Based on EEG Data)
Description: A responder is defined as a participant with a ≥50% reduction in seizure frequency from the baseline period of the previous study for LTFU participants. This OM was analyzed in participants <2 years (per EEG data) only.
Time Frame: as for outcome 6
Population: FAS: enrolled participants who had at least 1 dose of study drug in the study and had at least 1 completed post-baseline DRC or EEG. Overall number of participants analyzed consist of all participants (<2 years only [per EEG data]) evaluable for this OM. Per plan, participants were grouped per cohort linked to source (DRC for ≥2 years/EEG for <2 years) from which their seizure data is recorded.
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (BRV): Participants ≥1 Month to <2 Years
Number analyzed (Participants) | 8
percentage of participants | 75.0

9. Secondary Outcome: Absolute Change in Average Daily Frequency of POS in Participants <2 Years of Age With Typical Absence Seizures (Based on EEG Data)
Description: Absolute change in ADF is calculated as the baseline ADF minus post-baseline ADF. ADF is calculated as (number of seizures from central reader divided by stop date and time of EEG minus start date and time of EEG) multiplied to 60, multiplied to 24.
Time Frame: as for outcome 6
Population: Typical absence seizures data was not collected and analyzed.
Arm/Group | Brivaracetam (BRV): Participants ≥1 Month to <2 Years
Number analyzed (Participants) | 0

10. Secondary Outcome: Percent Change in Average Daily Frequency of POS in Participants <2 Years of Age With Typical Absence Seizures (Based on EEG Data)
Description: Percent change in average daily frequency (ADF) is calculated as absolute change in ADF divided by baseline ADF multiplied to 100. ADF is calculated as (number of seizures from central reader divided by stop date and time of EEG minus start date and time of EEG) multiplied to 60, multiplied to 24.
Time Frame: as for outcome 6
Population: Typical absence seizures data was not collected and analyzed.
Arm/Group | Brivaracetam (BRV): Participants ≥1 Month to <2 Years
Number analyzed (Participants) | 0

11. Secondary Outcome: 50% Responder Rate for Total Seizures (All Types) in Participants <2 Years of Age With Typical Absence Seizures (Based on EEG Data)
Description: A responder is defined as a participant with a ≥50% reduction in seizure frequency from the baseline period of the previous study for LTFU participants.
Time Frame: as for outcome 6
Population: Typical absence seizures data was not collected and analyzed.
Arm/Group | Brivaracetam (BRV): Participants ≥1 Month to <2 Years
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From Baseline to end of Study (up to 10 years)
Description: TEAEs are defined as AEs that had onset on or after the day of first BRV dose.
Arm/Group | Age Cohort: ≥1 Month to <2 Years | Age Cohort: ≥2 to <4 Years | Age Cohort: ≥4 to <12 Years | Age Cohort: ≥12 to <17 Years
All-Cause Mortality (participants affected / at risk) | 2/36 | 2/15 | 2/141 | 1/65
Serious Adverse Events (participants affected / at risk) | 14/36 | 8/15 | 42/141 | 19/65
Other Adverse Events (participants affected / at risk) | 30/36 | 13/15 | 120/141 | 51/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Cohort: ≥1 Month to <2 Years (N=36) | Age Cohort: ≥2 to <4 Years (N=15) | Age Cohort: ≥4 to <12 Years (N=141) | Age Cohort: ≥12 to <17 Years (N=65)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spina bifida (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth deposit (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 1 (1) | 3 (3) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (6) | 0 (0) | 4 (11) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurocysticercosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Greenstick fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iatrogenic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laparoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Underweight (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Astrocytoma, low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (6) | 1 (1) | 12 (20) | 2 (2)
Status epilepticus (Nervous system disorders) | 2 (3) | 0 (0) | 7 (12) | 2 (3)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 4 (7) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Complex partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Partial seizures with secondary generalisation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Simple partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural hygroma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anger (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal tubular acidosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrostomy (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Osteotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device extrusion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Cohort: ≥1 Month to <2 Years (N=36) | Age Cohort: ≥2 to <4 Years (N=15) | Age Cohort: ≥4 to <12 Years (N=141) | Age Cohort: ≥12 to <17 Years (N=65)
Anaemia (Blood and lymphatic system disorders) | 3 (5) | 0 (0) | 0 (0) | 1 (2)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 6 (6) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 6 (6) | 1 (1)
Strabismus (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypermetropia (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (19) | 5 (6) | 34 (61) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 7 (16) | 0 (0) | 21 (33) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0) | 12 (20) | 3 (9)
Constipation (Gastrointestinal disorders) | 7 (11) | 0 (0) | 10 (12) | 2 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 9 (10) | 8 (10)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 5 (5) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (6) | 1 (1) | 4 (5) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (21) | 1 (1) | 5 (5) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (5) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (3) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Teething (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (3) | 5 (6) | 6 (10)
Gait disturbance (General disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 15 (84) | 4 (11) | 37 (63) | 7 (9)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 10 (21) | 2 (9) | 39 (60) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 10 (19) | 5 (15) | 23 (38) | 8 (12)
Pharyngotonsillitis (Infections and infestations) | 5 (34) | 0 (0) | 21 (64) | 10 (20)
Gastroenteritis (Infections and infestations) | 8 (14) | 0 (0) | 16 (30) | 5 (6)
Influenza (Infections and infestations) | 5 (7) | 2 (2) | 16 (18) | 6 (6)
Bronchitis (Infections and infestations) | 7 (18) | 3 (11) | 16 (29) | 1 (1)
Rhinitis (Infections and infestations) | 5 (8) | 2 (3) | 16 (47) | 2 (6)
Nasopharyngitis (Infections and infestations) | 11 (44) | 4 (6) | 44 (114) | 16 (41)
Ear infection (Infections and infestations) | 2 (3) | 1 (2) | 10 (18) | 4 (4)
Tonsillitis (Infections and infestations) | 2 (2) | 1 (1) | 13 (21) | 2 (3)
Otitis media (Infections and infestations) | 4 (13) | 1 (1) | 10 (24) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 3 (3) | 6 (11) | 4 (5)
Varicella (Infections and infestations) | 4 (4) | 0 (0) | 9 (10) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 2 (3) | 0 (0) | 8 (9) | 2 (3)
Viral infection (Infections and infestations) | 3 (6) | 1 (1) | 7 (19) | 1 (2)
Conjunctivitis (Infections and infestations) | 5 (6) | 1 (2) | 4 (5) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (37) | 6 (11) | 1 (1)
Sinusitis (Infections and infestations) | 1 (3) | 2 (2) | 7 (12) | 1 (1)
Otitis media acute (Infections and infestations) | 3 (4) | 0 (0) | 4 (5) | 2 (2)
Pharyngitis bacterial (Infections and infestations) | 2 (3) | 0 (0) | 4 (4) | 1 (1)
Viral pharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (2) | 3 (3) | 0 (0)
Lice infestation (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 4 (16) | 9 (11) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (6) | 6 (10)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 6 (8) | 8 (11)
Weight decreased (Investigations) | 3 (3) | 0 (0) | 10 (13) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 6 (7) | 1 (1) | 16 (18) | 7 (8)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Underweight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 21 (58) | 16 (75)
Seizure (Nervous system disorders) | 3 (9) | 2 (2) | 17 (29) | 11 (17)
Somnolence (Nervous system disorders) | 3 (4) | 1 (1) | 15 (25) | 5 (5)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 7 (13) | 8 (16)
Complex partial seizures (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Muscle spasticity (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 5 (8) | 0 (0) | 14 (15) | 4 (4)
Aggression (Psychiatric disorders) | 0 (0) | 2 (2) | 14 (18) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3) | 3 (3) | 11 (14) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (4)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 4 (5) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (10) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 2 (4) | 19 (26) | 5 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 6 (7) | 5 (7)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0) | 10 (11) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 6 (8) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (18) | 0 (0) | 3 (4) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 10 (15) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT01364597/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT01364597/SAP_001.pdf